CLINICAL TRIAL: NCT04507828
Title: Combined Deep Inspiration Breath Hold (DIBH)-Expiration Planning Technique in Patients With Lung Tumors in Close Proximity to the Chest Wall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Lautenschlaeger, Assistant Professor of Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAON-IIR-IUSCC-0711
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: Radiation Treatment; Lung Cancer; Metastatic Cancer; Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined DIBH-Expiration Planning Technique (Experimental): Patients will undergo a 4D scan as well as a DIBH scan and an expiration breath hold scan. In order to develop a combined DIBH-Expiration treatment plan, the DIBH scan, the expiration phase of the 4D scan or the expiration breath hold scan will be used. If the radiation plan meets the coverage goals and normal tissue constraints, the patient will receive treatment using the new DIBH Planning Technique. If coverage and normal tissue constraints are not met per protocol, the patient will be treated per standard of care and not on protocol. Patients treated on protocol will undergo radiation treatment with SBRT for a total of 3 fractions and will receive each fraction no more frequently then every other day. Patients will then be evaluated at 1 month after SBRT completion and every 3 months for 2 years
  Interventions: Radiation: Treatment Planning using the DIBH Technique

INTERVENTIONS:
Radiation: Treatment Planning using the DIBH Technique — Different radiation plans will be generated-one using a DIBH scan with corresponding target and normal tissue contour and a second using an expiration scan with corresponding target and normal tissue contours. The expiration scan can be an expiratory gating scan averaging the expiratory breathing phases or an expiration breath hold scan as determined based on patient performance during simulation and relative tumor displacement compared to the DIBH scan. Then a third plan will be generated conceptually combining the two previous plans, named the DIBH-expiration composite plan.

SUMMARY:
The purpose of this study is to evaluate a new radiation planning and treatment delivery technique called Deep Inspiration Breath Hold (DIBH) and expiration technique. This technique will be used to treat patients who have tumors close to the chest wall and are candidates for Stereotactic Body Radiation Therapy (SBRT). This study will assess the reduction of radiation to the chest wall during treatment using this technique.

DETAILED DESCRIPTION:
Multiple studies have evaluated the efficacy of SBRT in patients with early stage lung cancer. The original Indiana University phase II trial evaluating three fraction SBRT with a total dose of 60-66 Gy for T1 and T2 (<7cm) lesions and median follow up of 50.2 months revealed a 3-year local failure rate of 5.7%. Tumor size and location did not impact tumor recurrence. [3]. RTOG 0236, which was a multi-institutional phase II trial evaluating the efficacy of three fraction SBRT for patients with peripherally located tumors, reported that 3-year local control rate was 98% with a median overall survival of 4 years and overall survival at 3 years of 56%. Long- term results of RTOG 0236 revealed a 5-year local failure rate of 7% and a 5-year overall survival rate of 40% [4, 5]. In addition, a pooled analysis of two randomized trials (Randomized study to Compare CyberKnife to Surgical Resection in Stage I Non-small Cell Lung Cancer [STARS] and the Trial of Either Surgery or Stereotactic Radiotherapy for Early Stage [IA] Lung Cancer [ROSEL]) comparing SBRT vs. lobectomy for operable stage I (T1-2aN0M0) NSCLC showed a 3-year overall survival for SBRT of 95% and for surgery of 79% (HR=0.14, p=0.037). There was no statistically significant difference between both groups in terms of 3-year rate of recurrence-free survival (HR = 0.69, p = 0.54) [5]. To evaluate the efficacy of SBRT (66 Gy in 3 fractions) compared to standard treatment (70 Gy in 35 fractions), 102 patients, with stage I inoperable NSCLC, were randomized to each treatment arm in the SPACE trial. The results were consistent with similar overall survival and progression free survival on both treatment groups. According to the TROG 09.02 CHISEL trial, stage I inoperable NSCLC patients treated with SBRT had superior local control of the primary disease (HR: 0.32) without an increase in major toxicity compared to patients treated with standard fractionation[6].

Pulmonary metastases frequently happen in patients with different types of cancer. Around 50% of patients who suffer from malignancy-related mortality have pulmonary metastasis at the time of autopsy [7]. In 1995, Hellman et al introduced the concept of oligometastases and the importance of aggressive surgical or ablative therapies to improve overall survival in this population [8]. As a result, SBRT technique has been widely used to treat pulmonary metastases. Multiple studies have evaluated this technique including a retrospective study evaluating 577 patients who undergo SBRT for pulmonary metastases that revealed 5-year local control of 46.3% and 5-year overall survival of 21.8% [9]. Based on the above findings, the researchers propose a prospective feasibility trial evaluating the combined DIBH-expiration planning and delivery technique in patients with lung tumors in close proximity to the chest wall who are candidates to receive lung SBRT per their standard care.

Based on the observed respiration dependent movement during CT simulation the study team will assign patients into two cohorts: A) Tumors with no overlap between respiratory states and B) Tumors with up to 50% overlap between respiratory states. For A, the study team will have a composite plan delivering half the dose using DIBH plan and the other half using the expiration phase plan for each fraction. For B) the radiation target will be subdivided into different zones with different zones receiving different prescriptions. The study plan will be compared to a standard plan specifically designed for the same patient. Researchers hypothesize that this technique will enable us to reduce chest wall V30 by 50% and deliver 54 Gy in 3 fractions while meeting all the dosimetric constraints. Cohorts A and B will be analyzed separately. Other dosimetric parameters will be evaluated in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 at time of consent
2. Karnofsky Performance Status (KPS) > 40
3. Ability to provide written informed consent and HIPAA authorization
4. Clinical or pathological diagnosis of primary lung cancer or metastasis to the lung
5. Tumors must be located within 2 cm from the chest wall, defined as the inner border of the 2-cm lung expansion volume (per TG101)
6. Plan to receive Lung SBRT

Exclusion Criteria:

1. Patients with tumors with > 50% overlap between respiratory states based on CT simulation will not be eligible for this study
2. Previous radiation therapy to the same site per investigator discretion
3. Inability to comply with treatment or standard of care follow up per investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Reduction in chest wall V30 using combined DIBH-expiration planning technique | 2 weeks (SBRT planning)
  The percentage of patients with an at least 50% reduction in chest wall V30 using combined DIBH-expiration planning technique in comparison to DIBH or expiration gating alone in the same patient

SECONDARY OUTCOMES:
Patients treated using DIBH planning technique | 8 weeks (treatment with SBRT)
  Percentage of patients treated with 54 Gy in 3 fractions using our new technique, who did not meet constraints for three fraction treatments using standard planning delivery techniques
Chest wall toxicity | 1 year
  Incidence of chest wall toxicity
Rib fracture | 1 year
  Incidence of rib fracture (based on surveillance imaging)
Local control rate | 2 year
  local control rates (defined as no tumor recurrence within 80% isodose line)
Time in treatment room | 8 weeks (completion of SBRT)
  Amount of on-table time in treatment room
Reduction in chest wall maximum dose | 2 weeks (SBRT planning)
  The calculated mean average of dosimetric reduction in chest wall maximum dose
Evaluate lung dose | 2 weeks
  Evaluation of mean lung dose

CONTACTS AND LOCATIONS:
Overall Officials: Tim Lautenschlager, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital / IU Simon Cancer Center, Indianapolis, Indiana, United States